CLINICAL TRIAL: NCT06088823
Title: Paresthesia in Hand and Antebrachium Following CardiacSurgery: Incidence, Risk Factors and Clinical Course
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Lind Jørgensen, Consultant, PhD, principal investigator, Rigshospitalet, Denmark
Other Study IDs: kandidatopgave NFL 2023
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Paresthesia; Peri-operative Injury; Complication,Postoperative; Upper Limb Nerve Lesion
Keywords: paresthesia upper limb; cardiac surgery; peri-operative complication
MeSH Terms: conditions — Paresthesia; Postoperative Complications | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No paresthesia: Patients that had no registration of post-operative paresthesia in hand or lower arm after cardiac surgery
  Interventions: Other: Heart surgery
- Paresthesia: Patients that had one o more registrations of post-operative paresthesia in hand or lower arm after cardiac surgery
  Interventions: Other: Heart surgery

INTERVENTIONS:
Other: Heart surgery — Adult cardiac surgery

SUMMARY:
To describe the incidence and severity of Paresthesia in Hand and Antebrachium in patients that have undergone CardiacSurgery.

DETAILED DESCRIPTION:
Some patients report tingling and/or numbness in hand and/or antebrachium after cardiac surgery, but potential risc factors and clinical course are not well described, and the incidence or severity is not known. Many factors may impact on the development of these complaints: age, BMI, pre-operative neurological deficits, diabetes, type, technique and duration of cardiac surgery, positioning of arms and hands during surgery, placement of the arterial line, time-to-extubation and post-operative positioning during this period.

The investigators aim to describe incidence and clinical course of these complaints and possibly identify modifiable risc factors in a retrospective cohort of patients that have undergone fast-track cardiac surgery, as a part of the on-going patient-centered quality improvement.

The study included 361 patients. Conclusion The incidence of hand paresthesia following cardiac surgery was 10%. This study found an increased occurrence of paresthesia after aortic valve surgery and prolonged aortic cross-clamp duration; these differences were not statistically significant. The impact of arterial line placement and patient positioning as a risk factor remains unclear. The majority of patients with paresthesia were overweight and had pre-existing comorbidity, with 11% reporting preoperative paresthesia. The clinical course of hand paresthesia following cardiac surgery was predominantly transient and not severe.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* cardiac surgery in the period from january 2022 to december 2023
* perioperative data entered into the quality database SafeBrain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients accepted for elective cardiac surgery, where peri-operative data have been entered in to the on-going quality databse SafeBrain (data protection journal number P-2020-27, Department of Healthcare law and dataprotection 1141, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen east, Denmark).
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of paresthesia in hand or lower arm after cardiac surgery | January 2022 - december 2023
  The number of patients with paresthesia in hand or lower arm after cardiac surgery, compared to total number of patients operated in the time period

SECONDARY OUTCOMES:
Risk factors for development og paresthesia in hand or lower arm after cardiac surgery | January 2022 - december 2023
  Analysis of the variables collected to identify possible risk factors for development og paresthesia in hand or lower arm after cardiac surgery
The clinical course of paresthesia in hand or lower arm after cardiac surgery | January 2022 - december 2023
  Qualitative description of the clinical course for paresthesia in hand or lower arm after cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Vibeke Renee Lind Jørgensen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No